CLINICAL TRIAL: NCT03167151
Title: A Parallel Group Phase I/II Marker Lesion Study to Assess the Safety, Tolerability and Efficacy of Intravenous or Intravesical Pembrolizumab in Intermediate Risk Recurrent Non-muscle Invasive Bladder Cancer
Brief Title: Pembrolizumab in Intermediate Risk Recurrent Non-muscle Invasive Bladder Cancer (NMIBC)
Acronym: PemBla
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study failed to recruit within the permitted timeframe
Sponsor: University of Oxford (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCTO-079; 2016-002267-33 (EudraCT Number)
Record Dates: First submitted 2017-05-02; First posted 2017-05-25 (Actual); Results first posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2019-12

CONDITIONS: Non-muscle Invasive Bladder Cancer (NMIBC)
Keywords: Recurrent intermediate risk NMIBC; Intravesical Pembrolizumab; Intravenous Pembrolizumab; Phase I/II; Marker-lesion; Non-muscle invasive bladder cancer (NMIBC)
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A Intravesical (Experimental): Intravesical Pembrolizumab (solution for infusion) 50-200 mg, given on D1, D8, D15, D22, D29, D36 & D64.
  Dose to be decided after safety run-in.
  Interventions: Drug: Pembrolizumab
- Arm B Intravenous (Active Comparator): Intravenous Pembrolizumab (solution for infusion), 200mg, given on D1, D22, D43, D64
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Solution for Infusion (Intravesical and Intravenous) 100mg/ 4ml vial
  Other Names: Keytruda

SUMMARY:
A parallel group, open label, multi-centre, phase I/II marker-lesion study of intravesical or intravenous pembrolizumab in recurrent intermediate risk NMIBC. Thirty patients (fifteen in each of two arms) will be randomised 1:1 to treatment with either intravesical pembrolizumab (Arm A) or intravenous pembrolizumab (Arm B). The main study will be preceded by a single institution safety run-in phase involving intra-patient dose escalation in six patients to confirm the safety and tolerability of intravesical pembrolizumab and the dose to be used in the randomised phase.

DETAILED DESCRIPTION:
Bladder cancer is the seventh most common cancer in the United Kingdom (UK) and ninth most common cancer worldwide. New strategies for treating this disease are urgently required to reduce recurrence and progression rates. Pembrolizumab is a type of immunotherapy drug that has been approved for use in certain types of melanoma and lung cancer. It is thought to work by helping the body's immune system to recognise and attack cancer. Drugs that work in a similar way have shown some encouraging results in studies treating patients with bladder cancer that has spread to other parts of the body, although they are not currently approved for treating either advanced or localised bladder cancer.

This trial is being performed to assess the safety and tolerability of giving pembrolizumab to patients with localised bladder cancer and to study what effects the drug has on the tumour; Participants will have all but one tumour (referred to as the marker lesion) removed during their transurethral resection of bladder tumour (TURBT) procedure at the start of the trial. After trial treatment, a further TURBT procedure will be carried out to remove the marker lesion, or if the marker lesion is no longer visible, a biopsy will be taken of the area where the growth was before.

After a safety run in with intra-patient dose escalation of intravesical pembrolizumab performed in paired patient cohorts, the trial will test two different ways of giving the pembrolizumab; directly into the bladder (intravesical) with 6 doses being received over 6 weeks and with a further dose approximately 3 weeks later, or into the blood stream via the veins (intravenous) with a dose being received every 3 weeks for a maximum of 4 doses.

36 eligible participants from across 3 UK centres will be randomly allocated to receive treatment by one of these ways. Following the end of treatment visit, patients will return to receiving standard care but receive follow-up for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the subject must:

1. Be willing and able to provide written informed consent for the trial and comply with the protocol scheduled follow-up visits and examinations for the duration of the study.
2. Be ≥ 18 years of age on day of signing informed consent.
3. Have recurrent NMIBC for which adjuvant treatment post TURBT would be a reasonable treatment option.
4. Main study only: a. Have recurrent, multiple (minimum 2) tumours consistent with NMIBC.

   b. Have at least one lesion of between 5-10mm in size clinically that can be left un-resected at TURBT as the marker lesion.

   c. Have histologically confirmed low grade transitional cell NMIBC at original and any subsequent diagnosis.
5. Have a normal upper urinary tract (as evidenced by ultrasound or CT urography within 2 years prior to randomisation) and no evidence of tumour in prostatic urethra at flexible cystoscopy.
6. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
7. Have adequate organ function as defined below:

   Haemoglobin (Hb) ≥ 9 g/dL without transfusion or erythropoietin (EPO) dependency Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L Total bilirubin ≤ 1.5 times the upper limit of normal (ULN) or direct bilirubin < ULN for subjects with total bilirubin levels > 1.5 x ULN Serum alanine aminotransferase (ALT) and/or serum aspartate aminotransferase (AST) ≤ 2.5 x ULN Serum creatinine OR Measured or calculated creatinine clearance ≤ 1.5 x ULN OR

   ≥ 60ml/min for subject with creatinine levels > 1.5 x institutional ULN Albumin ≥ 25g/L International Normalized Ratio (INR) or Prothrombin Time (PT) and Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or APTT is within therapeutic range of intended use of anticoagulants a Creatinine clearance should be calculated as per institutional standard
8. Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Both male and female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in section 5.1 for the course of the study and until 120 days after the last dose of the study medication.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Has received prior radiotherapy to the pelvis.
2. Has significant urinary incontinence or known bladder instability.
3. Main study only:

   1. Has more than 2 out of 3 of the following present at the current time: i. ≥8 tumours ii. Tumour ≥3cm in size iii. Frequent recurrence (>1/year)
   2. Has a previous history of any of the following: T1 tumour, high grade/G3 tumour, carcinoma in situ, multiple recurrent large (>3cm) Ta, G1 or G2 tumours.
   3. Had a primary tumour of unknown pathological stage or grade.
   4. Has disease for which resection of all visible tumours is not possible.
4. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 28 days of the first dose of trial treatment.
5. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Subjects requiring use of inhaled or intranasal corticosteroids or local steroid injections would not be excluded.
6. Has a known history of active tuberculosis (TB).
7. Has received intravesical Bacillus Calmette-Guerin (BCG) treatment within 30 days prior to the first dose of trial treatment.
8. Has hypersensitivity to pembrolizumab or any of its excipients.
9. Has had treatment with any other anti-cancer monoclonal antibody within 28 days prior to enrolment or who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
10. Has had treatment with prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks of administration of study drug or who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
11. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
12. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurological symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for a t least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin or physiologic corticosteroids replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
14. Has a known history of, or any evidence of active, non-infectious pneumonitis.
15. Has an active or intractable infection requiring systemic therapy.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
17. Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through to 120 days after the last dose of trial treatment.
19. Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed death ligand 1 (anti PD-L1), or anti-programmed death ligand 2 (anti-PD-L2) agent.
20. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
21. Has known active Hepatitis B (e.g. HBsAg reactive) or Hepatitis C (e.g. hepatitis C virus [HCV] RNA [qualitative] is detected).
22. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Protheroe, MRCP, FRCP, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (3):
- United Kingdom (3):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford, Surrey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initially, the plan was to recruit the 6 participants for the safety run-in phase of the study within 6 months. 9 patients, of which 6 were evaluable, were recruited at the Oxford Churchill Hospital site from 02 Mar 2018 until 31 Jan 2019. Due to the issues with slow recruitment, the steering committee decided to end recruitment on 31 Jan 2019
Pre-assignment Details: 9 participants were recruited onto the study. However, of the 9 participants, 2 were found to have no tumour present during their surgery and were therefore no longer eligible. A further 1 participant withdrew their consent after they had been recruited. Thus of 9 participants only 6 were eligible for analysis.
Groups:
- Safety run-in Phase Cohort 1: Cohort 1 in the safety run-in phase. Day 1 starting dose 50mg intravesical pembrolizumab
- Safety run-in Phase Cohort 2: Cohort 2 in the safety run-in phase. Day 1 starting dose 100mg intravesical pembrolizumab
- Safety run-in Phase Cohort 3: Cohort 3 in the safety run-in phase. Day 1 starting dose 200mg intravesical pembrolizumab
Period: Overall Study
Arm/Group | Safety run-in Phase Cohort 1 | Safety run-in Phase Cohort 2 | Safety run-in Phase Cohort 3
Started | 3 | 3 | 3
Completed | 2 | 2 | 2
Not Completed | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — No evidence of tumour at surgery | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety run-in Phase Cohort 1 | Safety run-in Phase Cohort 2 | Safety run-in Phase Cohort 3 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (0) | 66 (10.6) | 81 (7.8) | 73 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 2 | 1 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 2 | 2 | 2 | 6
Smoking status [Count of Participants; unit: Participants]
  Current | 0 | 1 | 0 | 1
  Ex-smoker | 2 | 1 | 1 | 4
  Never smoked | 0 | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Measure Description: ECOG performance status is a scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  Grade 0: fully active. Grade 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature Grade 2: up and about more than 50% of waking hours Grade 3: confined to bed or chair more than 50% of waking hours Grade 4: completely disabled Grade 5: dead
  Participants
    Performance Status 0 | 2 | 2 | 2 | 6
    Performance Status 1 | 0 | 0 | 0 | 0
Site of primary tumour [Count of Participants; unit: Participants]
  Bladder | 1 | 2 | 1 | 4
  Left renal pelvis | 0 | 0 | 1 | 1
  Urothelial | 1 | 0 | 0 | 1
Prior chemotherapy [Count of Participants; unit: Participants]
  Yes | 2 | 2 | 2 | 6
  No | 0 | 0 | 0 | 0
Prior surgery [Count of Participants; unit: Participants]
  Yes | 2 | 2 | 2 | 6
  No | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities (DLTs) to Assess the Safety, Tolerability and Toxicities of Intravesical Pembrolizumab After Transurethral Resection of Bladder Tumour (TURBT).
Description: Adverse events are categorised according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. Patients with intermediate risk Non-muscle Invasive Bladder Cancer (NMIBC) were assessed for dose limiting toxicity (DLT) and tolerability.
  Administration of at least 5 out of 6 treatments was required for the regime to be defined as tolerable.
Time Frame: Adverse event monitoring starts on the day of the TURBT procedure (Day -14) until 90 days post treatment, or 30 days following administration of the last dose of study medication if the subject initiates a new anticancer therapy.
Population: Six patients received at least 5 out of 6 scheduled treatments, or withdrew early due to drug-related toxicity, and hence these patients contributed to the DLT and tolerability analysis.
Measure: Number; unit: DLTs
Arm/Group | Safety run-in Phase Cohort 1 | Safety run-in Phase Cohort 2 | Safety run-in Phase Cohort 3
Number analyzed (Participants) | 2 | 2 | 2
DLTs | 0 | 0 | 0

2. Other Pre Specified Outcome: Correlation Between Expression of Programmed Death Ligand 1 (PD-L1) and Programmed Cell Death 1 (PD-1+) Infiltrating Lymphocytes and Efficacy of Pembrolizumab Therapy After TURBT.
Description: Pre treatment, during treatment (optional), and post treatment tumour samples Immunohistochemistry and Fluorescence-activated cell sorting (FACS) analysis to measure. Additionally, collection of an optional tumour sample at the time of recurrence or progression for research purposes will be performed if the patient provides consent for this. The optional tumour sample would be collected at the time of a standard care surveillance cystoscopy or resection if the patient had a repeat TURBT in standard care.
Time Frame: Day -14 TURBT, optional Day 50 TURBT, Day 85 TURBT and where applicable optional follow-up period ≤ 24 months
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Definition of Gene Expression Signatures and Genetic Profiles Capable of Predicting Efficacy of Pembrolizumab Treatment in NMIBC Patients.
Description: Gene expression profiling and DNA sequencing on pre-treatment blood and tumour samples to predict efficacy of pembrolizumab treatment in NMIBC patients.
Time Frame: Day 1 pre-treatment
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Analysis of T-cell Receptor (TCR) Repertoire and Clonality of Infiltrating T-cells in Resected Tumour Specimens, Urine and Normal Bladder Tissue.
Description: Evaluating the effects of pembrolizumab treatment on the immunological profile and tumour specific immune responses in patients with intermediate risk NMIBC.
Time Frame: Day 1 to 92
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Analysis of TCR Repertoire and Clonality of Peripheral Blood Mononuclear Cells (PBMC) Before, During and After Treatment.
Description: Identification of myeloid or T cell responses in the tumour microenvironment associated with the response to treatment with pembrolizumab.
Time Frame: Day 1 to 92
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Analysis of Cytokines in Blood and Urine.
Description: Identification of myeloid or T cell responses in the tumour microenvironment associated with response to treatment
Time Frame: Day 1 to 92
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event monitoring starts on the day of the TURBT procedure (Day -14) until 90 days post treatment, or 30 days following administration of the last dose of study medication if the subject initiates a new anticancer therapy.
Description: The investigator monitored each patient for clinical and laboratory evidence of adverse events on a routine basis throughout the study.
Arm/Group | Safety run-in Phase Cohort 1 | Safety run-in Phase Cohort 2 | Safety run-in Phase Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety run-in Phase Cohort 1 (N=2) | Safety run-in Phase Cohort 2 (N=2) | Safety run-in Phase Cohort 3 (N=2)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety run-in Phase Cohort 1 (N=2) | Safety run-in Phase Cohort 2 (N=2) | Safety run-in Phase Cohort 3 (N=2)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flushes (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Rash over bilateral shins
Rigors (General disorders) | 1 (1) | 0 (0) | 0 (0)
Urgency-Frequency Syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (3)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the issues with slow recruitment, the decision was taken to end the trial after the safety run in phase, before the randomised phase began.

This meant only a very small number of patients could be analysed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT03167151/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT03167151/SAP_001.pdf